CLINICAL TRIAL: NCT01486719
Title: Sensory Reconstruction of Finger Pulp Defect Using a Dorsal Digital Island Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other); The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHEN-19750306
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Trauma
Keywords: Finger pulp reconstruction; dorsal branch; proper digital nerve; palmar arterial arch; dorsal digital island flap
MeSH Terms: conditions — Wounds and Injuries | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Sensate Dorsal Digital Island Flap — This article reports repair of the finger pulp defect using the dorsal digital island flap. Both dorsal branches of the proper digital nerves (PDNs) were used for maximal sensory restoration.
  Other Names: Surgical Flap; Island Flap

SUMMARY:
Sensory reconstruction of the finger pulp is a challenging problem. This article reports repair of the finger pulp defect using the dorsal digital island flap. Both dorsal branches of the proper digital nerves (PDNs) were used for maximal sensory restoration.

DETAILED DESCRIPTION:
From February 2008 to May 2009, the flap harvested from the dorsum of the middle phalanx of the same finger was used in 12 fingers in 12 patients. The flaps ranged in size from 2.0 × 2.0 cm to 2.8 × 2.2 cm. The mean pedicle length was 1.2 cm. Neurorrhaphy between the dorsal branches of the PDN and PDN was performed in both sides in all cases. Sensibility of the reconstructed finger pulp was evaluated by static 2-point discrimination (2PD) and Semmes-Weinstein monofilament test. The range of motion of the donor fingers was measured. The data were compared to those of the opposite sides.

ELIGIBILITY:
Inclusion Criteria:

1. a finger pulp defect > 1.5 cm in length
2. necessity to preserve finger length
3. patients younger than 60 years .

Exclusion Criteria:

1. injury to the dorsum of the middle phalanx of the reconstructed finger that precluded its use as donor site
2. injury to the course of the vascular pedicle or opposite PDA
3. defects < 1.5 cm in length.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination test | Patients were followed for 16-23 months (mean, 19 months)
  The patients were assessed at follow-up by an independent senior surgeon who did not attend the treatments. Evaluation included active range of motion (ROM) of the DIP and proximal interphalangeal (PIP ) joints, and static 2-point discrimination (2PD) and Semmes-Weinstein monofilament test of the reconstructed finger pulps. These measurements were compared with those on the contralateral site. According to the Michigan Hand Outcomes Questionnaire (MHQ), patients reported their satisfaction with the appearance of the injured hand. The questions based on a 5-point response scale.

SECONDARY OUTCOMES:
Semmes-Weinstein monofilament test | Patients were followed for 16-23 months (mean, 19 months)
  The patients were assessed at follow-up by an independent senior surgeon who did not attend the treatments. Evaluation included active range of motion (ROM) of the DIP and proximal interphalangeal (PIP ) joints, and static 2-point discrimination (2PD) and Semmes-Weinstein monofilament test of the reconstructed finger pulps. These measurements were compared with those on the contralateral site.

REFERENCES:
- [Result] Bene MD, Petrolati M, Raimondi P, Tremolada C, Muset A. Reverse dorsal digital island flap. Plast Reconstr Surg. 1994 Mar;93(3):552-7. PMID 8115510
- [Result] Pelissier P, Casoli V, Bakhach J, Martin D, Baudet J. Reverse dorsal digital and metacarpal flaps: a review of 27 cases. Plast Reconstr Surg. 1999 Jan;103(1):159-65. doi: 10.1097/00006534-199901000-00025. PMID 9915177
- [Derived] Chen C, Tang P, Zhang X. Sensory reconstruction of a finger pulp defect using a dorsal homodigital island flap. Plast Reconstr Surg. 2012 Nov;130(5):1077-1086. doi: 10.1097/PRS.0b013e318267ef99. PMID 22777035